CLINICAL TRIAL: NCT04300517
Title: The Effect of Protein Supplement on Paraspinal Muscles in Patients Undergoing Lumbar Posterior Spine Fusion Surgery
Brief Title: Effect of Protein Supplement on Paraspinal Muscles in Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University (Other)
Responsible Party: Principal Investigator, Zahra Vahdat Shariatpanahi, Principal Investigator, Shahid Beheshti University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1398/802
Record Dates: First submitted 2020-03-03; First posted 2020-03-09 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Spine Surgery
Keywords: Protein supplement; Spine Surgery; Paraspinal Muscles

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- protein supplement (Experimental): Intervention patients will be received protein diet (1.2 g/kg/day) and protein supplement (36 g/day) for 1 month after surgery.
  Interventions: Drug: Three sachet of protein supplement to be mixed in with water used daily
- maltodextrin (Placebo Comparator): Control patients will be received protein diet (1.2 g/kg/day) and maltodextrin for 1 month after surgery.
  Interventions: Drug: Three sachet of protein supplement to be mixed in with water used daily

INTERVENTIONS:
Drug: Three sachet of protein supplement to be mixed in with water used daily — Three sachet of protein supplement to be mixed in with water used daily
  Other Names: Pure-protein®

SUMMARY:
Protein intake in spinal fusion surgery can prevent paraspinal muscle atrophy by maintaining muscle mass, regeneration, and growth. Also, by reducing the amount of pseudarthrosis, pain and disability can have a positive effect on recovery.

The high prevalence of this type of surgery, the instability and degeneration of adjacent surfaces of fused sections, lumbar muscle atrophy, increased muscle tissue fat, and negative impact on patient recovery, also with regard to the fact that research has so far aimed to determine The effect of protein supplementation on para-spinal muscles has not been studied in patients undergoing posterior lumbar spine fusion surgery, therefore clinical trials are necessary. In this trial patients undergoing elective posterior spine fusion surgery are divided into two groups of intervention or control.

DETAILED DESCRIPTION:
A randomized, double blind, controlled trial will be conducted in patients undergoing elective posterior spine fusion surgery in Tehran, Iran. After a full review of the inclusion and exclusion criteria and explanation of the risks and benefits of the study, written consent form will be completed. The participants are 80 eligible posterior spine fusion surgery patients, aged ≥ 18 years. Intervention patients will be received 36 grams of protein supplement along with diet containing 1.2 g/kg/day of protein for 30 days after surgery and control patients will be received maltodextrin along with diet containing 1.2 g/kg/day of protein 30 days after surgery. Patients will be evaluated for occurrence of paraspinal muscles after 3 months surgery

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18-65 years
* Body mass index 18.5-30
* Candidate for the elective posterior spine fusion
* Without history of severe liver disorder
* Without history of Kidney disorder
* Without history of diabetes
* Without history of trauma and fracture of the vertebral
* Without history of osteoporosis
* Without history of Gastrointestinal malabsorption
* Without history of Parathyroid gland disorders
* Without taking medications that affect the metabolism of bone, such as calcitonin, bisphosphonate, corticosteroid
* No smoking
* Without history of neuromuscular diseases such as dystrophies and neurological disorders

Exclusion Criteria:

* Allergy or intolerance to protein or maltodextrine supplement
* Unwillingness to continue cooperation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
The thickness of the paraspinal muscles in CT scan | 3 months after surgery
  The thickness of the paraspinal muscles (multifidus, erector spinae, Quadratus, and Lumborum) in CT scan

SECONDARY OUTCOMES:
Degree and severity of paraspinal muscle mass atrophy in CT scan | baseline, and 3 months after surgery
  Degree and severity of paraspinal muscle mass atrophy (multifidus, erector spinae, Quadratus, and Lumborum) in CT scan

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nutrition and Food Technology, Shahid Beheshti University of Medical Sciences, Shohada Tajrish Hospital, Tehran, Iran